CLINICAL TRIAL: NCT03513302
Title: Dietary Nitrate and Muscle Power With Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Andrew Coggan, Associate Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1712579448
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Aging; Sarcopenia
Keywords: nitric oxide
MeSH Terms: conditions — Sarcopenia | interventions — Nitrates

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo
- nitrate (Active Comparator)
  Interventions: Dietary Supplement: nitrate

INTERVENTIONS:
Dietary Supplement: placebo — 2 x 70 mL concentrated beet root juice depleted of nitrate per day for 14 days.
  Other Names: Beet It Sport Nitrate 400 placebo
  Arms: placebo
Dietary Supplement: nitrate — 2 x 70 mL concentrated beet root juice per day for 14 days.
  Other Names: Beet It Sport Nitrate 400
  Arms: nitrate

SUMMARY:
The purpose of this study is to see if drinking beetroot juice (BRJ) is beneficial for aging patients. We hope to determine the effect of BRJ on exercise performance. BRJ improves exercise performance in athletes and normal people. We are trying to determine if BRJ improves exercise performance in aging patients. We will be comparing the effects of BRJ versus the effects of a placebo (BRJ without the nitrates that are naturally occurring in beets and other similar foods). It is thought that the benefits of BRJ may come from its natural nitrate content. Although BRJ is available for purchase in grocery stores, for the purposes of this study it is considered investigational, which means that it has not been approved as a medical therapy.

DETAILED DESCRIPTION:
This study consists of two parts separated by a 14 day wash-out. Subjects will be randomly assigned to receive either the BRJ or placebo during the first part. During the second part they will receive the opposite of what they had during the first part. This is considered a double-blind study, which means neither the subjects nor the investigators will know what form (BRJ or placebo) a subject is receives.

Study Visit One (Screening) 1-2 hours

The purpose of the screening visit is to explain all aspects of the study. It will also determine if subjects can participate in the study. Subjects will provide a complete medical history and undergo a physical exam. They will have their blood drawn (about 1.5 teaspoons) and provide a urine sample. They will also practice the entire neuromuscular function exercise test. During this test, the strength of their muscles will be determined by having them kick, push and/or pull back as hard as you can while their leg is strapped to an exercise device. A vital signs monitor will measure your blood pressure, heart rate, and rhythm.

During the remainder of the study subjects will be instructed to consume their normal diet. However, they will be asked to avoid eating foods high in nitrate such as beets, spinach, and collard greens the evening before each visit. They will be asked to refrain from the use of antibacterial mouthwash, such as Listerine or Cepacol, during the study. Chewing gum, alcohol, and food and drinks containing caffeine (coffee, tea, chocolate, and soft drinks) should be avoided 24 hours prior to each visit. They will be asked to fast for 12 hour prior to each study visit.

Study Visit Two - Approximately 5 hours

At the beginning of this visit a catheter (small, flexible, sterile plastic tube) will be placed through a vein in one of the subject's arms. This is for collection of blood samples. Blood will be drawn four times during this visit. Each draw will be 6 mL or about 1.2 teaspoons. The first blood draw will check nitrate and nitrite levels. They will then have a breath test to check nitric oxide. They will then drink 140 mL (about 2/3 of a cup) of BRJ (or placebo). Blood and breath samples will be obtained every hour. Heart rate and blood pressure will be measured at the same times the blood and breath samples are obtained. Subjects will then rest quietly in a private room for about 2 hours after ingestion of BRJ (or placebo) then will perform:

* The neuromuscular function test that was practiced during the screening visit.
* After completing the exercise test they will undergo a muscle biopsy of their thigh muscle. First, the area will be sterilized and numbed with an injection. Next, a small incision (about ¼ inch) will be made and a small biopsy needle will be used to collect a small sample of your muscle (about the size of a pencil eraser). This will be performed on the leg opposite of that used during the neuromuscular test.
* One final blood and breath sample will then be obtained.
* Subjects will then be provided a 7 day supply of BRJ (or placebo) and will continue to drink two bottles (about 5 oz) every morning.
* Subjects will also be provided with an activity tracker. This will be worn at the hip during all waking hours except when bathing or swimming. This monitor will measure total activity time and sedentary time.

Study Visit Three - 1-2 hours

Subjects will return to the research center with the empty BRJ bottles. At this visit a single blood (1.2 teaspoon) and breath sample will be collected. Subjects will then complete a questionnaire to rate how tired they felt during the previous week. They will be provided another 7 day supply of BRJ (or placebo) and will continue to drink two bottles every morning.

Study Visit Four - Approximately 5 hours Subjects will return to the research center and undergo the same procedures as they did in Study Visit Two. They will also complete a questionnaire that will rate how tired they felt during the previous week.

Washout After visit four subjects will undergo a 14 day washout period where they will not drink the BRJ (or placebo). There are no dietary restrictions at this time; subjects may consume caffeine, alcohol, gum, mouthwash, etc. Subjects will then repeat Study Visits Two, Three, and Four again. However, during this they will be given the opposite form of BRJ you had received before.

Study Visit Five Subjects will repeat the procedures completed during Study Visit Two.

Study Visit Six Subjects will repeat the procedures completed during Study Visit Three.

Study Visit Seven Subjects will repeat the procedures completed during Study Visit Four.

ELIGIBILITY:
Inclusion Criteria:

In good health, as determined by the investigator's review of history (provided by subject at screening visit), physical examination, and routine blood and urine tests (done at screening visit)

Exclusion Criteria:

Men and women <65 or >79 years of age

* Unable to provide informed consent
* Currently pregnant or lactating (given the age range for the study, verbal confirmation by subject is believed to be sufficient)
* Current smokers
* Significant orthopedic limitations or other contraindications to strenuous exercise
* Those taking phosphodiesterase inhibitors (e.g., Viagra)
* Those taking proton pump inhibitors, antacids, xanthine oxidase inhibitors, or on hormone replacement therapy
* Those taking anti-coagulants (e.g., Coumadin) or on anti-platelet therapy
* History of neuromuscular disease (e.g., cervical spondylotic radiculomyelpathy, lumbar spondylosis, amyotrophic lateral sclerosis, Guillain-Barré syndrome, and acquired demyelinating polyneuropathies), cardiovascular disease (e.g., > stage I hypertension, heart failure, myocardial infarction/ischemia, significant myocardial or pericardial diseases (e.g. amyloidosis, constriction), moderate or severe valvular disease, renal disease, liver disease, or anemia

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Coggan, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Health and Human Sciences, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coggan AR. Dietary Nitrate and Muscle Function in Humans: Acute versus Chronic Mechanisms. Med Sci Sports Exerc. 2018 Apr;50(4):874. doi: 10.1249/MSS.0000000000001489. No abstract available. PMID 29547495
- [Background] Coggan AR, Broadstreet SR, Mikhalkova D, Bole I, Leibowitz JL, Kadkhodayan A, Park S, Thomas DP, Thies D, Peterson LR. Dietary nitrate-induced increases in human muscle power: high versus low responders. Physiol Rep. 2018 Jan;6(2):e13575. doi: 10.14814/phy2.13575. PMID 29368802
- [Background] Coggan AR, Broadstreet SR, Mahmood K, Mikhalkova D, Madigan M, Bole I, Park S, Leibowitz JL, Kadkhodayan A, Thomas DP, Thies D, Peterson LR. Dietary Nitrate Increases VO2peak and Performance but Does Not Alter Ventilation or Efficiency in Patients With Heart Failure With Reduced Ejection Fraction. J Card Fail. 2018 Feb;24(2):65-73. doi: 10.1016/j.cardfail.2017.09.004. Epub 2017 Sep 12. PMID 28916479
- [Background] Coggan AR, Peterson LR. Dietary Nitrate and Skeletal Muscle Contractile Function in Heart Failure. Curr Heart Fail Rep. 2016 Aug;13(4):158-65. doi: 10.1007/s11897-016-0293-9. PMID 27271563
- [Background] Rimer EG, Peterson LR, Coggan AR, Martin JC. Increase in Maximal Cycling Power With Acute Dietary Nitrate Supplementation. Int J Sports Physiol Perform. 2016 Sep;11(6):715-720. doi: 10.1123/ijspp.2015-0533. Epub 2016 Aug 24. PMID 26641379
- [Background] Coggan AR, Leibowitz JL, Spearie CA, Kadkhodayan A, Thomas DP, Ramamurthy S, Mahmood K, Park S, Waller S, Farmer M, Peterson LR. Acute Dietary Nitrate Intake Improves Muscle Contractile Function in Patients With Heart Failure: A Double-Blind, Placebo-Controlled, Randomized Trial. Circ Heart Fail. 2015 Sep;8(5):914-20. doi: 10.1161/CIRCHEARTFAILURE.115.002141. Epub 2015 Jul 15. PMID 26179185
- [Background] Coggan AR, Leibowitz JL, Kadkhodayan A, Thomas DP, Ramamurthy S, Spearie CA, Waller S, Farmer M, Peterson LR. Effect of acute dietary nitrate intake on maximal knee extensor speed and power in healthy men and women. Nitric Oxide. 2015 Aug 1;48:16-21. doi: 10.1016/j.niox.2014.08.014. Epub 2014 Sep 6. PMID 25199856

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Nitrate: Placebo (2 x 70 mL concentrated beet root juice depleted of nitrate per day) for 14 days, 14 day washout, Nitrate (2 x 70 mL concentrated beet root juice containing nitrate per day) for 14 days
- Nitrate Then Placebo: Nitrate (2 x 70 mL concentrated beet root juice containing nitrate per day) for 14 days, 14 day washout, placebo (2 x 70 mL concentrated beet root juice depleted of nitrate per day) for 14 days
Period: First Intervention (14 Days)
Arm/Group | Placebo Then Nitrate | Nitrate Then Placebo
Started | 23 | 24
Completed | 8 | 8
Not Completed | 15 | 16
Not completed — Screen failure | 15 | 16
Period: Washout (14 Days)
Arm/Group | Placebo Then Nitrate | Nitrate Then Placebo
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention (14 Days)
Arm/Group | Placebo Then Nitrate | Nitrate Then Placebo
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximal Knee Extension Velocity
Description: *Maximal* knee extension velocity was determined by having participants perform knee extensions at velocities of 0, 1.57, 3.14, 4.57, and 6.14 radians per second on an isokinetic dynamometer (device that controls velocity while measuring torque). Peak power at each velocity was calculated by multiplying the measured torque by that velocity, then a parabolic function was fit to these calculated data to predict *maximal* knee extensor velocity. Higher values are better.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: radians per second
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 16 | 16
radians per second | 12.2 (1.9) | 12.7 (2.1)

2. Primary Outcome: Muscle Knee Extensor Power
Description: This outcome was determined by having participants perform knee extensions at velocities of 0, 1.57, 3.14, 4.57, and 6.14 radians per second on an isokinetic dynamometer (device that controls velocity while measuring torque). *Peak* power at each velocity was calculated by multiplying the measured torque by that velocity, then a parabolic function was fit to these calculated data to predict *maximal* knee extensor power. Higher values are better.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Watts per kilogram body mass
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 16 | 16
Watts per kilogram body mass | 3.98 (1.18) | 4.26 (1.37)

3. Primary Outcome: Maximal Knee Extension Velocity
Description: *Maximal* knee extension velocity was determined by having participants perform knee extensions at velocities of 0, 1.57, 3.14, 4.57, and 6.14 rad/s on an isokinetic dynamometer (device that controls velocity while measuring torque). Peak power at each velocity was calculated by multiplying the measured torque by that velocity, then *maximal* knee extensor velocity was determined by fitting a parabolic function to these data (*maximal* knee extension velocity = 2 x fitted velocity at which *maximal* power is developed). Higher values are better.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: rad/s
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 16 | 16
rad/s | 12.2 (1.8) | 12.7 (1.8)

4. Primary Outcome: Maximal Knee Extension Power
Description: *Maximal* knee extension power was determined by having participants perform knee extensions at velocities of 0, 1.57, 3.14, 4.57, and 6.14 rad/s on an isokinetic dynamometer (device that controls velocity while measuring torque). *Peak* power at each velocity was calculated by multiplying the measured torque by that velocity, then *maximal* power was determined by fitting a parabolic function to these data. Higher values are better.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: W/kg
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 16 | 16
W/kg | 4.23 (1.21) | 4.31 (1.26)

5. Other Pre Specified Outcome: Plasma Nitrate
Description: Plasma nitrate concentrations were measured using high performance liquid chromatography.
Time Frame: 0,1,2,3 hours after treatment at 1 day
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 16 | 16
umol/L
  0 h | 35 (24) | 39 (19)
  1 h | 35 (22) | 601 (258)
  2 h | 33 (20) | 698 (214)
  3 h | 33 (16) | 661 (247)

6. Other Pre Specified Outcome: Plasma Nitrate
Description: Plasma nitrate concentrations
Time Frame: 0,1,2,3 hours after treatment at 14 days
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 16 | 16
umol/L
  0 h | 37 (20) | 190 (153)
  1 h | 35 (13) | 740 (241)
  2 h | 35 (11) | 815 (281)
  3 h | 35 (14) | 780 (292)

7. Other Pre Specified Outcome: Plasma Nitrite
Description: Plasma nitrite concentrations were measured using high performance liquid chromatography.
Time Frame: 0,1,2,3 hours after treatment at 1 day
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 16 | 16
umol/L
  0 h | 0.364 (0.283) | 0.400 (0.356)
  1 h | 0.382 (0.338) | 0.904 (0.826)
  2 h | 0.379 (0.401) | 1.104 (0.847)
  3 h | 0.374 (0.376) | 1.243 (1.078)

8. Other Pre Specified Outcome: Plasma Nitrite
Description: Plasma nitrite concentrations were measured using high performance liquid chromatography.
Time Frame: 0,1,2,3 hours after treatment at 14 days
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 16 | 16
umol/L
  0 h | 0.307 (0.294) | 0.615 (0.671)
  1 h | 0.308 (0.247) | 0.972 (1.039)
  2 h | 0.353 (0.344) | 1.053 (1.144)
  3 h | 0.275 (0.286) | 0.989 (1.039)

9. Other Pre Specified Outcome: Perceived Fatigue
Description: Patient-Reported Outcomes Measurement Information System perceived fatigue questionnaire (PROMIS 8a). Results given as T-score with mean of 50 and standard deviation of 10. Lower is better.
Time Frame: 1 and 14 days of treatment
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 16 | 16
T-score
  1 d | 42.3 (9.1) | 43.2 (8.9)
  14 d | 39.3 (7.1) | 40.8 (6.6)

10. Other Pre Specified Outcome: Physical Function
Description: Patient-Reported Outcomes Measurement Information System physical function questionnaire (PROMIS 20a). Results given as T-score with mean of 50 and standard deviation of 10. Higher is better.
Time Frame: 1,14 days of treatment
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 16 | 16
T-score
  1 day | 53.0 (6.8) | 52.2 (7.4)
  14 days | 54.7 (6.8) | 57.0 (6.3)

11. Post Hoc Outcome: Plasma 8-hydroxydeoxyguanosine
Description: Plasma 8-hydroxydeoxyguanosine is an indicator of oxidative damage to DNA/RNA. It was measured using a commercial enzyme-linked immunosuppressant assay kit. Lower is better.
Time Frame: 1 and 14 days of treatment
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 16 | 16
mg/mL
  Pre-treatment | 11.4 (4.0) | 11.5 (4.5)
  Post-treatment | 11.6 (3.9) | 11.7 (4.5)

12. Post Hoc Outcome: Plasma Protein Carbonyls
Description: Protein carbonyls are an indicator of oxidative damage to proteins. It was measured using a commercial enzyme-linked immunosuppressant assay kit. Lower is better.
Time Frame: 1 and 14 days of treatment
Measure: Mean (Standard Deviation); unit: nmol/mg
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 16 | 16
nmol/mg
  Pre-treatment | 3.71 (1.40) | 4.00 (1.67)
  Post-treatment | 3.79 (1.67) | 4.46 (2.17)

13. Post Hoc Outcome: Plasma 4-hydroxynonenal
Description: 4-hydroxynonenal is an indicator of oxidative damage to lipids (fats). It was measured using a commercial enzyme-linked immunosuppressant assay kit. Lower is better.
Time Frame: 1 and 14 days of treatment
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 16 | 16
ug/mL
  Pre-treatment | 43.9 (25.0) | 38.1 (24.6)
  Post-treatment | 38.4 (26.6) | 35.7 (24.0)

ADVERSE EVENTS:
Time Frame: 14 days of first intervention + 14 days of washout + 14 days of second intervention
Description: *IN KEEPING WITH INSTITUTIONAL POLICIES, ALL INDIVIDUALS ENROLLED IN (CONSENTED FOR) THE STUDY WERE CONSIDERED "AT RISK", EVEN IF THEY DID NOT PASS SCREENING AND DID NOT RECEIVE THE INTERVENTION.*
Groups:
- Screening Period: Adverse events during screening, prior to arm/group assignment
- Placebo: Placebo (2 x 70 mL concentrated beet root juice depleted of nitrate per day) for 14 days
- Nitrate: Nitrate (2 x 70 mL concentrated beet root juice containing nitrate per day) for 14 days
Arm/Group | Screening Period | Placebo | Nitrate
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 27/47 | 5/16 | 4/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screening Period (N=47) | Placebo (N=16) | Nitrate (N=16)
Abnormal laboratory finding (Metabolism and nutrition disorders) | 9 (18) | 0 (0) | 0 (0)
Abnormal laboratory finding (Endocrine disorders) | 8 (10) | 0 (0) | 0 (0)
Abnormal laboratory finding (Blood and lymphatic system disorders) | 16 (33) | 0 (0) | 0 (0)
Abnormal laboratory finding (Renal and urinary disorders) | 7 (7) | 0 (0) | 0 (0)
Abnormal laboratory finding (Hepatobiliary disorders) | 5 (5) | 0 (0) | 0 (0)
Toothache (General disorders) | 0 (0) | 1 (1) | 0 (0) — Toothache
Muscle soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea/diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epidermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
High blood pressure (Cardiac disorders) | 14 (14) | 3 (4) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT03513302/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT03513302/ICF_001.pdf